CLINICAL TRIAL: NCT01177735
Title: Phase II Trial of Pomalidomide in GEP-defined High-risk Multiple Myeloma That is Relapsing or Refractory to Prior Therapy
Brief Title: Pomalidomide in Gene Expression Profiling (GEP)-Defined High-risk Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113385; UARK 2010-01 (Other: UAMS); NCT01426503 (obsolete NCT alias)
Record Dates: First submitted 2010-05-14; First posted 2010-08-09 (Estimated); Results first posted 2015-03-04 (Estimated); Last update posted 2021-04-22 (Actual); Status verified 2017-10

CONDITIONS: Multiple Myeloma
Keywords: Pomalidomide; multiple myeloma; relapsed
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pomalidomide (Experimental)
  Interventions: Drug: Pomalidomide

INTERVENTIONS:
Drug: Pomalidomide — Only enough CC-4047 for 1 cycle of therapy may be provided to the patient each cycle. Participants will receive CC-4047 4 mg/day for 21 days, every 28 days. Treatment will continue until disease recurrence or untoward toxicity.
  Other Names: CC-4047

SUMMARY:
This is a phase II study, open-label, single institution trial of pomalidomide in GEP-defined, high-risk relapsing/refractory multiple myeloma. Prior therapy must have included lenalidomide. Patient accrual is 30 over a 2 year period.

Primary objective:

* To determine progression-free survival (PFS) after initiation of pomalidomide therapy

Secondary objective:

* To determine the response rate (CR, n-CR, VGPR) and duration of response after pomalidomide therapy.
* To determine gene expression profiling (GEP) changes exerted within 48 hours of initiation of daily pomalidomide dosing.
* To determine gene expression profiling (GEP) changes exerted within 48 hours of initiation 3 concurrent days of exposure to lenalidomide.
* To determine MRI- and PET-CT-defined CR in studies obtained at baseline and every 6 month examinations.

DETAILED DESCRIPTION:
Pomalidomide is a 2nd generation immunomodulatory agent (IMiD®) with greater efficacy than lenalidomide and with a similar toxicity spectrum. Phase I trials have shown that pomalidomide 1 to 5 mg is well-tolerated1,2.

TT3 has been remarkably successful in the management of newly diagnosed MM, inducing CR rates of >60% and 4-year estimates of overall and event-free survival of 85% and 75%. Of those achieving CR, estimated 4-year CR rate is 85%. TT3 maintenance has been with either VTD in 2003-33 or VRD in 2006-66, so that pomalidomide's role in overcoming refractoriness to lenalidomide can be assessed.

Pharmacogenomic investigations comparing GEP data obtained at baseline and 48hr post-treatment have been performed in case of thalidomide, dexamethasone, lenalidomide, bortezomib and melphalan3. Thus, as most patients on TT3 had baseline and 48-hr GEP investigations performed after bortezomib, the opportunity exists to investigate, at the time of relapse, not only a re-challenge with bortezomib with 48hr GEP but also pomalidomide's effect.

This is a phase II study, open-label, single institution trial of pomalidomide in GEP-defined, high-risk relapsing/refractory multiple myeloma. Prior therapy must have included lenalidomide.

ELIGIBILITY:
Inclusion Criteria:

* Participant has multiple myeloma, relapsed or resistant to prior therapy.
* Participant has high-risk disease, as defined by any of the following:

  * GEP risk score of > 0.66 OR
  * Metaphase based abnormalities of 1q or 1p OR
  * LDH > 360 U/L
* Participant has received prior therapy with lenalidomide-containing regimen and has been determined to be refractory, resistant, or relapsed.
* Participant has no significant peripheral neuropathy (< grade 3 by the most current NCI CTCAE version)
* Participant has adequate hematopoietic reserve as defined by platelet count ≥ 50,000/µL and ANC of > 1000/µL.
* Participant has adequate renal function as defined by serum creatinine < 2 mg/dL.
* Participant has adequate hepatic function, defined by serum Total bilirubin </= 1.5 mg/dL and AST (SGOT) and ALT (SGPT) </= x ULN.
* Participant is 18 years of age or greater.
* Participant has not received anti-cancer therapy within 4 weeks prior to treatment on this study.
* Zubrod ≤ 2, unless solely due to symptoms of MM-related bone disease.
* Disease free of prior malignancies for >/= 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix or breast.
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours prior to starting lenalidomide or CC-4047 and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide or CC-4047.
* All patients must be informed of the investigational nature of this study and must sign and give written voluntary consent in accordance with institutional and federal guidelines.
* Willing and able to take aspirin or alternate prophylactic anticoagulation.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or breast feeding females.
* Men unwilling to use a condom (even if they have undergone a prior vasectomy) while having intercourse with any woman, while taking the drug and for 4 weeks after stopping treatment.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 28 days of baseline.
* Known hypersensitivity to lenalidomide.
* The development of erythema nodosum if characterized by a desquamating rash while taking lenalidomide, CC-4047 or similar drugs.
* Any prior use of CC-4047.
* Concurrent use of other anti-cancer agents or treatments.
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible.
* Active malignancy (exception of non melanoma skin cancer or in situ cervical or breast cancer).
* Active DVT or PE that has not been therapeutically anticoagulated.
* ≥ grade 3 peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saad Usmani, MD, Principal Investigator — University of Arkansas for Medical Sciences, Myeloma Institute for Research and Therapy
Locations (1):
- University of Arkansas for Medical Sciences, Myeloma Institute for Research and Therapy, Little Rock, Arkansas, United States

REFERENCES:
- See also: Myeloma Institute for Research and Therapy at The University of Arkansas for Medical Sciences — http://myeloma.uams.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pomalidomide
Started | 71
Completed | 0
Not Completed | 71

BASELINE CHARACTERISTICS:
Arm/Group | Pomalidomide
Number analyzed (Participants) | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.25 (76.161)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 43
Region of Enrollment [Number; unit: participants]
  United States | 71

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) After Initiation of Pomalidomide Therapy
Description: Progression -free survival (PFS) after initiation of pomalidomide therapy. Progressive disease is defined as increase of > 25% from lowest response value in any one or more of the following: Serum M-component and/or (the absolute increase must be > 0.5 g/dL); Urine M-component and/or (the absolute increase must be > 200 mg/24 h); Only in patients without measurable serum and urine M-protein levels; the difference between involved and uninvolved FLC levels. The absolute increase must be > 10 mg/dL; Bone marrow plasma cell percentage; the absolute percentage must be > 10%; Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; Development of hypercalcaemia (corrected serum calcium > 11.5 mg/dL or 2.65 mmol/L) that can be attributed solely to the plasma cell proliferative disorder.
Time Frame: 1 year following initiation of pomalidomide therapy
Measure: Number; unit: percentage of participants
Arm/Group | Pomalidomide
Number analyzed (Participants) | 71
percentage of participants | 13

ADVERSE EVENTS:
Arm/Group | Pomalidomide
Serious Adverse Events (participants affected / at risk) | 6/71
Other Adverse Events (participants affected / at risk) | 71/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pomalidomide (N=71)
Acute renal failure (Renal and urinary disorders) | 2 (2)
Hospitalization for sinus infection (Infections and infestations) | 1 (1)
Hospialization for progressive disease, sepsis and pneumonia (Infections and infestations) | 3 (3)
Hospitalization for removal of port (Injury, poisoning and procedural complications) | 1 (1)
Hospitalization for fever (Infections and infestations) | 1 (1)
RSV Pneumonia (Infections and infestations) | 2 (2)
Fever neutropenia dehydration (Infections and infestations) | 1 (1)
Hospitalization for neutropenic fever (Infections and infestations) | 4 (4)
Hospitalization due to acute liver failure hepatitis B flare (Infections and infestations) | 1 (1)
Hospitalization for pneumonia (Infections and infestations) | 1 (1)
Atrial Fibrilation (Cardiac disorders) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Hypoxia (General disorders) | 1 (1)
Hospitalization dyspnea due to congestive heart failure (Cardiac disorders) | 1 (1)
Hospitalization for shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea on exertion (Cardiac disorders) | 1 (1)
Hospitalization for bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Blood and lymphatic system disorders) | 1 (1)
Hospitalization for hypotension (Cardiac disorders) | 2 (2)
Respiratory failure secondary to opioid overdose (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalization for intractable pain, low fever (Nervous system disorders) | 1 (1)
Hospitalization for acute respiratory distress syndrome, encephalopathy, fatigue (Nervous system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Intrahepatic chemotherapy (Surgical and medical procedures) | 1 (1)
Paraparesis, spinal cord compression (Nervous system disorders) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1)
Fracture of T7 with possible cord compression (Injury, poisoning and procedural complications) | 1 (1)
Deep vein thrombosis and cerebrovascular accident (Cardiac disorders) | 1 (1)
Blood transfusion (Blood and lymphatic system disorders) | 1 (1)
Wrong dosage dispensed (Surgical and medical procedures) | 1 (1)
Hospitalization with fever and low blood pressure (Cardiac disorders) | 1 (1)
Acute diarrhea (Gastrointestinal disorders) | 1 (1)
Hospitalization for Pneumonia and gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Hospitalization for diarrhea and dizziness (Gastrointestinal disorders) | 1 (1)
Elevated liver function test (Infections and infestations) | 1 (1)
Deep vein thrombosis diagnosis (Vascular disorders) | 1 (1)
Hospitalization for sepsis (Infections and infestations) | 1 (1)
Worsening renal failure (Renal and urinary disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Pneumonia, fever and altered mental status (Infections and infestations) | 1 (1)
Severe cough, shortness of breath and hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of breath fever chills (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalization for parainfluenza type 2 (Infections and infestations) | 1 (1)
Mental status changes and bacteremia (Psychiatric disorders) | 1 (1)
Recurrent multifocal pneumonia (Infections and infestations) | 1 (1)
Upper respiratory infection and fever (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute onset diarrhea and acute renal insufficiency (Infections and infestations) | 1 (1)
Hospitalization due to transient ischemic attack (Vascular disorders) | 1 (1)
Shortness of breath with wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Recurrent bilateral pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pomalidomide (N=71)
Leukopenia (Blood and lymphatic system disorders) | 71
Thrombocytopenia (Blood and lymphatic system disorders) | 71
Anemia (Blood and lymphatic system disorders) | 71
Blood/Bone Marrow (General disorders) | 71 — For some "Other" (non-serious) adverse events, only the affected organ system was recorded/reported.
Cardiac Arrhythmia (Cardiac disorders) | 7
Cardiac General (Cardiac disorders) | 12 — For some "Other" (non-serious) adverse events, only the affected organ system was recorded/reported.
Constitutional Symptoms (General disorders) | 55
Dermatology / Skin (Skin and subcutaneous tissue disorders) | 31 — For some "Other" (non-serious) adverse events, only the affected organ system was recorded/reported.
Gastrointestinal (Gastrointestinal disorders) | 44 — For some "Other" (non-serious) adverse events, only the affected organ system was recorded/reported.
Hemorrhage / Bleeding (Injury, poisoning and procedural complications) | 8
Hepatobiliary / Pancreas (Hepatobiliary disorders) | 70 — For some "Other" (non-serious) adverse events, only the affected organ system was recorded/reported.
Infection (Infections and infestations) | 29
Lymphatics (Blood and lymphatic system disorders) | 10 — For some "Other" (non-serious) adverse events, only the affected organ system was recorded/reported.
Metabolic/Laboratory (Metabolism and nutrition disorders) | 66 — For some "Other" (non-serious) adverse events, only the affected organ system was recorded/reported.
Musculoskeletal / Soft Tissue (Musculoskeletal and connective tissue disorders) | 24 — For some "Other" (non-serious) adverse events, only the affected organ system was recorded/reported.
Neurology (Nervous system disorders) | 55 — For some "Other" (non-serious) adverse events, only the affected organ system was recorded/reported.
Ocular / Vision (Eye disorders) | 6 — For some "Other" (non-serious) adverse events, only the affected organ system was recorded/reported.
Pain (General disorders) | 40
Pulmonary / Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 40 — For some "Other" (non-serious) adverse events, only the affected organ system was recorded/reported.
Renal / Genitourinary (Renal and urinary disorders) | 45 — For some "Other" (non-serious) adverse events, only the affected organ system was recorded/reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes